CLINICAL TRIAL: NCT05933408
Title: Is Triggering Receptor Expressed On Myeloid Cells 1 (TREM-1) Protein a New Marker of Serious Infectious Complications in Colorectal Surgery? - Case-matched Pilot Study
Brief Title: TREM-1 - a New Marker of Serious Infectious Complications in Colorectal Surgery?
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Karolina Zawadzka, Medical Doctor, Principal Investigator, Jagiellonian University
Other Study IDs: TREM-1
Record Dates: First submitted 2023-06-28; First posted 2023-07-06 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Colorectal (Colon or Rectal) Cancer
Keywords: colorectal; cancer; complications; infectious; TREM-1; marker
MeSH Terms: conditions — Colonic Neoplasms; Neoplasms; Communicable Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with serious infectious complications: Complications were graded according to the five grade Clavien-Dindo classification (CD 1-5). Complications have been divided into mild (CD 1-2) and severe (CD 3-5).
  Interventions: Diagnostic Test: TREM-1
- Patients without complications: Patients with infectious complications who formed group 1, were matched 1:1 with patients without complications (group 2). Case-matched analysis was performed by selecting patients for the control group from the group of patients paired by age, ASA scale, stage of cancer and type of surgery.

INTERVENTIONS:
Diagnostic Test: TREM-1 — The TREM-1 (triggering receptor expressed on myeloid cells-1) glycoprotein is a receptor involved in the activation of monocytes and neutrophils during the inflammatory process. There are many reports indicating the soluble form of this receptor is a reliable diagnostic marker of infection and inflammatory response induced by trauma. Therefore the investigators aimed to investigate the potential use of soluble TREM-1 to predict serious infectious complications in patients undergoing laparoscopic colorectal surgery.Blood samples were drawn four times: on the day of surgery (preoperatively) and on the three following postoperative days (PODs).
  Groups: Patients with serious infectious complications

SUMMARY:
The aim of this study is to investigate the potential use of soluble TREM-1 (sTREM-1) to predict serious infectious complications in patients undergoing laparoscopic colorectal surgery. Patients with colon or rectal cancer, who underwent elective laparoscopic colorectal cancer surgery between November 2018 and February 2020 were included into study. Blood samples for the TREM-1 protein assay were collected from each patient four times: preoperatively and on three following postoperative days (PODs).

Patients with infectious complications who formed group 1, were matched 1:1 with patients without complications (group 2). Case-matched analysis was performed by selecting patients for the control group from the group of patients paired by age, ASA scale, stage of cancer and type of surgery.

DETAILED DESCRIPTION:
The TREM-1 (triggering receptor expressed on myeloid cells-1) glycoprotein, which belongs to the immunoglobulin superfamily, is a receptor involved in the activation of monocytes and neutrophils during the inflammatory process. There are many reports indicating the soluble form of this receptor is a reliable diagnostic marker of infection and inflammatory response induced by trauma [9, 10]. TREM-1 has been described as a mean to assess the risk of the occurrence of infections in some surgical conditions, but no one has studied its application in predicting complications in patients who underwent elective laparoscopic resection of colorectal cancer [11, 12]. Therefore, the investigators set out to investigate the potential use of soluble TREM-1 (sTREM-1) to predict serious infectious complications in patients undergoing laparoscopic colorectal surgery.

Patients with colon or rectal cancer, who underwent elective laparoscopic colorectal cancer surgery between November 2018 and February 2020 were included into study. Blood samples for the TREM-1 protein assay were collected from each patient four times: preoperatively and on three following postoperative days (PODs).

Clinical data and demographic information of patients (age, sex, comorbidities, ASA (American Society of Anaesthesiologists) physical status) were prospectively collected on database. After the surgery, the database was supplemented with data related to the procedure (type of surgery, operative time, intraoperative blood loss) and treatment results (complication, length of hospital stay (LOS)).

Patients with infectious complications who formed group 1, were matched 1:1 with patients without complications (group 2). Case-matched analysis was performed by selecting patients for the control group from the group of patients paired by age, ASA scale, stage of cancer and type of surgery.

Complications were graded according to the five grade Clavien-Dindo classification (CD 1-5). Complications have been divided into mild (CD 1-2) and severe (CD 3-5).

Since 2012, in our department the perioperative care of all patients is carried out based on the ERAS protocol and laparoscopic approach has been the gold standard in colorectal surgery at our center.

ELIGIBILITY:
Inclusion Criteria:

- adult patients (>18 y/o) with histopathologically confirmed colorectal adenocarcinoma who underwent laparoscopic resection of the colon and/or rectum

Exclusion Criteria:

* open or emergency surgery,
* multivisceral resection
* stage IV cancer according to American Joint Committee on Cancer (AJCC) classification system
* concomitant inflammatory bowel disease
* autoimmune systemic disease
* other active infection
* when conversion to open resection was necessary

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with infectious complications who formed group 1, were matched 1:1 with patients without complications (group 2). Case-matched analysis was performed by selecting patients for the control group from the group of patients paired by age, ASA scale, stage of cancer and type of surgery.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
TREM-1 levels on the first postoperative day | first postoperative day
  TREM-1 levels on the first day after surgery in patients with and without infectious complications

SECONDARY OUTCOMES:
TREM-1 levels on the second postoperative day | second postoperative day
  TREM-1 levels on the second day after surgery in patients with and without infectious complications
TREM-1 levels on the third postoperative day | third postoperative day
  TREM-1 levels on the third day after surgery in patients with and without infectious complications

CONTACTS AND LOCATIONS:
Locations (1):
- Jagiellonian University Medical College, Krakow, Małopolska, Poland

IPD SHARING:
Plan to Share IPD: No